CLINICAL TRIAL: NCT07130136
Title: Post-Market Clinical Follow-Up of the Osia System and Evaluation of Benefits of Transitioning From the Baha Connect System to the Osia System in Adult Bone Conduction Implant Recipients With Mixed or Conductive Hearing Loss
Brief Title: Post-market Evaluation of the Transition From the Baha Connect System to the Osia System in Adult Bone Conduction Implant Recipients
Acronym: OSIRIS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear (Industry)
Collaborators: TFS HealthScience (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLTD5858
Record Dates: First submitted 2025-08-12; First posted 2025-08-19 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-07

CONDITIONS: Bone Conduction; Hearing Loss, Conductive; Hearing Loss, Mixed
Keywords: Bone Conduction; Speech perception; Patient satisfaction
MeSH Terms: conditions — Hearing Loss, Conductive; Hearing Loss, Mixed Conductive-Sensorineural; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: Within-group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cochlear™ Osia® System and Cochlear™ Baha® System (Experimental): Participants undergoing transition from the Baha Connect System to the Osia System will complete a series of assessments and questionnaires designed to evaluate the clinical performance and user satisfaction of both systems.
  Interventions: Device: Cochlear™ Osia® System; Device: Cochlear™ Baha® System

INTERVENTIONS:
Device: Cochlear™ Osia® System — The Osia System consists of the OSI300 Implant, Osia 2 Sound Processor, Osia 2 Sound Processor Magnets, Osia 2 Sound Processor Magnet Tool, Osia Fitting Software 2 (OFS 2), and Osia Smart App.
Device: Cochlear™ Baha® System — The Baha Connect System consists of the BIA300 (BI300 Implant and BA300 Abutment), Baha 7 Sound Processor, and Baha Fitting Software 7 (BFS 7).

SUMMARY:
The goal of this interventional study is to confirm the safety and performance of the latest generation Osia System and to examine its benefits compared to the Baha Connect System in adults with mixed or conductive hearing loss who have a pre-existing Baha implant and Abutment (BIA300) and are transitioning to the Osia System.

The main questions this study aims to answer are:

* Is the safety and performance of the Osia System confirmed by study findings?
* What are the benefits of the Osia System compared to the Baha Connect System?

Participants will:

* Undergo speech performance testing in both quiet and noisy environments
* Provide ratings for various questionnaires

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Implanted with a Cochlear Baha BI300 Implant in combination with a Cochlear Baha BA300 Abutment (Baha Connect)
* Mixed or conductive hearing loss in the ear implanted with the Baha Connect System
* Bone conduction thresholds with pure tone average (PTA4; mean of 0.5, 1, 2, and 4 kHz) of ≤ 55 dB HL in the ear implanted with the Baha Connect System
* Experience of at least 6 months with the Baha Connect System
* Candidate is judged by the investigator to be dissatisfied with their current Baha Connect System due to medical issues, e.g., recurrent adverse skin reactions, and is considered likely to benefit from transitioning to an Osia System
* Candidate is a fluent speaker in the language used to assess speech perception performance
* Candidate is willing and able to provide written informed consent
* Candidate has a retrospective medical record from the time of implantation with the Baha Connect System which the investigational site is authorized to review

Exclusion Criteria:

* Candidate with single-sided deafness (air conduction thresholds with pure tone average (PTA4; mean of 0.5, 1, 2 and 3 kHz) of ≤ 20 dB HL in the good ear)
* Candidate with an acute infection (Holgers grade 4) at the implant site at the time of screening
* Unable or unwilling to comply with the requirements of the clinical investigation as determined by the Investigator
* Investigator site personnel directly affiliated with this study and/or their immediate families; immediate family is defined as a spouse, parent, child, or sibling
* Cochlear employees or employees of Contract Research Organizations or contractors engaged by Cochlear for the purposes of this investigation
* Current participation, or participation in another interventional clinical study/trial in the past 30 days, involving an investigational drug or device (unless Cochlear sponsored and determined by the investigator or Sponsor to not impact this investigation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2028-11 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change (within-subject) in speech reception threshold in noise measured at 65 dB SPL (pre-operative unaided and post-operative aided with the Osia System) | At Baseline Visit 2 (2-3 weeks after Baseline Visit 1) and at 3-months post-implantation (Day 90)
  Speech perception in noise will be assessed using the Bamford-Kowal-Bench-Speech in Noise (BKB-SIN) test, which assesses speech recognition in the presence of background noise. This test consists of lists of sentences, each containing 3-4 key words, presented at 65 dB SPL with increasingly progressive levels of background noise. One point is awarded for each correctly repeated word, and the results are used to calculate the signal-to-noise ratio (SNR) at which 50% of the key words (SNR-50) are correctly repeated.

SECONDARY OUTCOMES:
The incidence rates of Adverse Events (AEs) and Device Deficiencies (DD) (both systems) | From screening through to the end of study at 6 months (Day 180), including any additional visits (Ad Hoc)
  The incidence rates of all reported AEs per device type and specific rates for DD will be assessed. A breakdown by category will be provided to indicate the proportion of patients experiencing each category (by severity, by relatedness to device or procedure, and by seriousness) of AE and DD.
The frequency and types of healthcare interventions related (both systems) | At Baseline Visit 1 (2-3 weeks prior to Baseline Visit 2) to study end (Day 180)
  The frequency and types of healthcare interventions (e.g., follow-up visits, treatments, and hospitalisations) associated with the use of the device systems will be collected.
Change (within-subject) in word recognition score in quiet measured at 65 dB SPL (pre-operative unaided and post-operative aided with the Osia System) | At Baseline Visit 2 (2-3 weeks after Baseline Visit 1) and at 3 months post-implantation (Day 90)
  Word recognition in quiet will be measured using the Arthur Boothroyd (AB) Speech Test, which assesses speech recognition in a quiet surrounding. The AB test involves monosyllables presented at 65 dB SPL, with scores recorded as the percentage of correctly repeated words at each presentation level.
Total score and attribute scores from the Health Utilities Index (HUI)-2/3 questionnaire (Osia System) | At Baseline Visit 2 (2-3 weeks after Baseline Visit 1) and at 3 months post-implantation (Day 90)
  The HUI-2/3 perception-based questionnaire involves a comprehensive health status and health-related quality of life, using 15 questions comprised of 8 attributes: Vision, Hearing, Speech, Ambulation, Dexterity, Emotion, Cognition, and Pain. A score is given that reflects overall quality of life, where 1 means perfect health and 0 means a state equivalent to death.
Global score and subscale scores from the Speech Spatial Qualities of Hearing Scale (SSQ-49) questionnaire (Osia System) | At Baseline Visit 2 (2-3 weeks after Baseline Visit 1) and at 3 months post-implantation (Day 90)
  The SSQ-49 involves a self-reported hearing function and the impact of hearing treatment in daily life across a variety of listening situations. It includes 3 subcategories: Speech Hearing, Spatial Hearing, and Qualities of Hearing, with each question rated on a Likert scale from 0-10 (minimum - maximum hearing abilities).
Change (within-subject) in global Satisfaction with Amplification in Daily Life (SADL) score and subscale scores (both systems) | At Baseline Visit 2 (2-3 weeks after Baseline Visit 1) and at 3 months post-implantation (Day 90)
  The SADL involves a self-report inventory to quantify satisfaction with hearing aids. It consists of 15 items, a generated global satisfaction score, and 4 subscale scores (positive effect, service & cost, negative features, and personal image). The scores range from 1 to 7, where the higher scores indicate greater satisfaction with the hearing device.
Change (within-subject) in word recognition score in quiet measured at 65 dB SPL (both systems) | At Baseline Visit 2 (2-3 weeks after Baseline Visit 1) and at 3 months post-implantation (Day 90)
  Word recognition in quiet will be measured using the Arthur Boothroyd (AB) Speech Test, which assesses speech recognition in a quiet surrounding. The AB test involves monosyllables presented at 65 dB SPL, with scores recorded as the percentage of correctly repeated words at each presentation level.
Change (within-subject) in word recognition score in quiet measured at 50 dB SPL (both systems) | At Baseline Visit 2 (2-3 weeks after Baseline Visit 1) and at 3 months post-implantation (Day 90)
  Word recognition in quiet will be measured using the Arthur Boothroyd (AB) Speech Test, which assesses speech recognition in a quiet surrounding. The AB test involves monosyllables presented at 50 dB SPL, with scores recorded as the percentage of correctly repeated words at each presentation level.
Change (within-subject) in word recognition score in quiet measured at 80 dB SPL (both systems) | At Baseline Visit 2 (2-3 weeks after Baseline Visit 1) and at 3 months post-implantation (Day 90)
  Word recognition in quiet will be measured using the Arthur Boothroyd (AB) Speech Test, which assesses speech recognition in a quiet surrounding. The AB test involves monosyllables presented at 80 dB SPL, with scores recorded as the percentage of correctly repeated words at each presentation level.

CONTACTS AND LOCATIONS:
Overall Officials: PRS Specialist, Study Director — Cochlear Ltd
Locations (3):
- United Kingdom (3):
  - Royal National Ear, Nose and Throat and Eastman Dental Hospitals, London
  - Nottingham Auditory Implant Programme, Nottingham
  - Sheffield Teaching Hospitals, Sheffield

IPD SHARING:
Plan to Share IPD: No
Cochlear do not have an approved platform for public sharing of IPD collected in this study. Data may be provided to individual researchers on request.